CLINICAL TRIAL: NCT02573662
Title: Metabolic Complications Following Knee Injury in Young and Middle Aged Patients
Acronym: OrthoMetKnee
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haugaard, Steen Bendix, M.D., DMSc (Individual)
Collaborators: Hölmich, Per, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: AH-ORTHOMET-01
Record Dates: First submitted 2015-03-13; First posted 2015-10-12 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Glucose Metabolism Disorders; Lipid Metabolism Disorders; Sedentary Lifestyle
Keywords: Metabolic complications; Type 2 diabetes; Sedentary lifestyle; Low grade inflammation; Lipid metabolism; Glucose metabolism; Bone metabolism; Physical inactivity
MeSH Terms: conditions — Glucose Metabolism Disorders; Lipid Metabolism Disorders; Sedentary Behavior; Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection; Absorptiometry, Photon; Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine sampling
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case subjects: Physical active non-diabetic individuals of age 18 to 50 years, who are undergoing knee surgical procedures at the Arthroscopic Center at Amager/Hvidovre Hospitals are recruited as cases for this case-control study. OGTT, blood- and urine sampling and DXA scans will be performed 3 times throughout the study period.
  Interventions: Biological: Blood and Urine sampling; Radiation: DXA scan; Biological: OGTT
- Control group: Non-diabetic individuals matched for age, gender and physical activity are recruited as control subjects to establish a reference level likely to image the cases before they experienced their knee injury. Blood- and urine sampling, OGTT and DXA scans will be carried out 1-3 times for each control subject. No lifestyle intervention is implemented.
  Interventions: Biological: Blood and Urine sampling; Radiation: DXA scan; Biological: OGTT

INTERVENTIONS:
Biological: Blood and Urine sampling — Blood and Urine Sampling
Radiation: DXA scan — Scan of Lumbar columna and neck of femur/hip Scan of visceral/subcutaneous fatty tissue
Biological: OGTT — Oral Glucose Tolerance Test for Minimal Model analysis for insulin sensitivity and Lipid oxidation

SUMMARY:
Introduction This study evaluates the effect on glucose, lipid and bone metabolism following knee orthopedic procedures in healthy and physically active individuals. The sedentary rehabilitation period following these procedures may impact negatively on glucose, lipid and bone metabolic pathways, whereas the more physically active rehabilitation period instituted 6 weeks after surgery is hypothesized to impact positively.

Perspective This study will establish whether the well-known effects on glucose, lipid and bone metabolism of a sedentary lifestyle can be observed already following 6 weeks of physical inactivity in otherwise healthy and physically fit young and middle aged individuals. Investigators will thereby add knowledge to previous findings following strict bed-rest in healthy individuals on glucose, lipid and bone metabolism. In a clinical perspective it is important to examine the extent to which healthy individuals deteriorate in various metabolic pathways to better understand the pathophysiology behind these defects both in healthy individuals and in patients, who undergo bed rest or an equal reduction in physical activity as part of their rehabilitation.

Study design 16 physical active non-diabetic individuals of age 18 - 50 years who are undergoing knee surgical procedures at the Arthroscopic Center at Amager/Hvidovre Hospitals are recruited as cases for this case-control study.

10 non-diabetic control subjects matched for age, gender and physical activity are recruited to establish a reference level.

* The individuals will bring in morning spot urine for measurement of soluble urokinase plasminogen activating receptor (suPAR), creatinine, albumin and orosomucoid. Weight and height and waist and hip circumference will be measured.
* Oral glucose tolerance test (OGTT) with ingestion of 75 g glucose during 5 min from baseline (0 min). Plasma for glucose, insulin, C-peptide, non-esterified fatty acid (NEFA) will be drawn
* Before OGTT blood will be drawn for measurement of HbA1c, total cholesterol, LDL, HDL, triglyceride, Na, K, creatinine, hemoglobin (HgB), C-reactive protein (CRP), leukocytes, alanintransaminase (ALAT), alkaline phosphatase, Ca++, D vitamin, TSH, bone turnover markers (BTM), suPAR, interleukin 6 (IL6), TNFa, high-sensitivity C-reactive protein (hsCRP), lipid density profiling and lipid particle size.
* Dual energy X-ray absorptiometry (DXA) of hip, lumbar columna, visceral and subcutaneous fat is measured by Hologic Discovery scanner.

DETAILED DESCRIPTION:
Hypothesis Implementation of a sedentary lifestyle with almost no physical activity in otherwise physical active individuals undergoing knee orthopaedic surgical procedures will during 6 weeks (4 to 8 weeks)

* derange insulin sensitivity and glucose effectiveness
* decrease disposition index
* imply hyper-secretion of incretin hormones and glucagon
* compensatory decrease in insulin clearance
* decrease lipid oxidation
* increase visceral adipose tissue
* increase number of low density lipoprotein particles and a decrease the particle size
* increase immune and low grade inflammatory response as measured in plasma and urine
* induce bone loss in hip as measured by bone mineral density (BMD)
* increase bone resorption and decrease bone formation as measured by selected bone turnover markers.

The proposed negative changes in bone, lipid and glucose metabolism are thought to reverse at least partly so, during active physical rehabilitation during week 6 through week 16.

Statistics Ten days of bed rest in 13 healthy young individuals showed a 20% (P<0.05) significant decrease in insulin sensitivity and a 50% (P<0.05) reduction in lipid oxidation. Thirty-one days of bed rest in 8 healthy women was significantly associated with bone loss in total hip (2.07%, P<0.001).

As the present study does not imply strict bed rest but exhibit a longer sedentary period of following up as the above studies and include a larger number of participants we are very likely to exhibit a power > 80% at significance level

Ethical issues The study is approved by the local scientific ethical committee and the Danish Data Protection Agency. The study adheres to the Danish Act on Processing of Personal Data and, Danish Act on Health and the Helsinki II convention of clinical trials. The study will be announced at the clinicaltrials.gov homepage. All participants are informed about the purpose of the study, all ethical issues and a written consent is obtained before participation.

Personal data from patient medical files will be accessed by principal investigator to gather information concerning the knee injuries in order to identify and characterize the knee injury for each subject. Personal data concerning demographic relations such as gender and age will be accessed as well to ensure the case subjects meet the inclusion criteria and for statistically use. To make assessments on study participation, the principal investigator will also gain access to relevant data from the patient s medical files concerning illnesses or conditions the case subject might report. The X-ray radiation from 1 DXA scan equals 1 day of background radiation in Denmark. Thus 3 DXA scans throughout the study period are equal to 3 days of background radiation. This amount of radiation is 30-fold less than that of a single standard CT-scan of abdomen. In other words the dose of radiation is so low that a calculation of risk is not possible.

The amount of blood drawn during the approximately 16 weeks of participation in the study is less than 500 ml, which is the standard amount of blood drawn at a single donation of blood from a blood donor. The use of intravenous cannula can cause irritation or infection of vein or insertion site. All procedures will be performed as described in SOP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of age 18 to 50 years
* Physically active >/= 1.5 hours/week up till baseline examination
* Physically active at least 2.5 hours/week before knee injury.
* The participants should undergo one of the following orthopaedic surgical procedures; Medial patella-femoral ligament (MPFL) surgery, Anterior Crusiate Ligament (ACL) and/or Posterior Crusiate Ligament (PCL) surgery, Knee Cartilage Injury surgery
* Informed written consent

Exclusion Criteria:

* BMI >/= 30 kg/m2
* Not physically active before surgical procedure as measured by questionnaire
* Known diabetes mellitus or HbA1c >/= 48 mol/mol
* Clinical significant anemia, liver or kidney disease as judged by the sponsor or principal investigator.
* Thyroid function abnormality (TSH < 0.1 or TSH > 10)
* Calcium metabolic derangement, Ca++ < 1.1 or Ca++ > 1.40
* Known osteoporosis

Inclusion/exclusion criteria for control subjects are similar except from surgical procedure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixteen physical active non-diabetic individuals of age 18 to 50 years who are undergoing knee surgical procedures at the Arthroscopic Center at Amager/Hvidovre Hospitals are recruited as cases for this case-control study.
  Ten non-diabetic individuals matched for age, gender and physical activity are recruited as control subjects.
  The pre-surgical physical activity level is expected to be lower than their habitual physical activity, however more than that which would be expected from individuals with a sedentary life-style.
  At least 6 of the control subjects will be examined another two times, that is, after 6 weeks and after 16 weeks for the purpose of time controls.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Baseline to week 6
  Glucose metabolic: -insulin sensitivity as measured by MinModel-OGTT

SECONDARY OUTCOMES:
Change in glucose metabolism | Baseline to week 6 and to week 16
  * Change in beta-cell responsiveness compared to insulin sensitivity (disposition index)
  * Change in glucose effectiveness
  * Change in insulin clearance
  * Change in visceral adipose tissue
  * Change in incretin secretion compared to insulin resistance and insulin secretion
Lipid metabolism | Baseline to week 6 and to week 16
  * Change ind lipid oxidation as measured by MinModel-NEFA
  * Change in lipolysis
  * Change in rates of which NEFA leaves plasma pool
Bone Metabolism | Baseline to week 6 and to week 16
  * BMD changes in total hip; changes in total BMD
  * change in lumbar BMD
  * changes in BTM of bone resorption (CTX) and formation (P1NP)
Atherosclerotic markers | Baseline to week 6 and to week 16
  * change in low and high density lipoprotein particles and in particle size
  * changes in TNFa, IL6, hsCRP, suPAR and orosomucoid
Change in insulin sensitivity | week 6 and to week 16
  Glucose metabolic: -insulin sensitivity as measured by MinModel-OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Per Hölmich, MD, DMSc, Principal Investigator — Amager Hospital
Locations (1):
- Amager University Hospital, Copenhagen, Denmark